CLINICAL TRIAL: NCT07401589
Title: Association of Postoperative SpO₂/FiO₂ Ratio With Body Mass Index, STOP-BANG Score, and Analgesic Methods in Patients Undergoing Laparoscopic Surgery in Reverse Trendelenburg Position
Brief Title: Postoperative SpO₂/FiO₂ Ratio and Analgesic Methods in Laparoscopic Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, ass. prof, Istinye University
Other Study IDs: 293-2025
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Hypoxemia
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative Observational Cohort
  Interventions: Other: Standard of Care
- control
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — No intervention is applied in this study. Patients are managed according to routine clinical practice. Demographic data, body mass index, STOP-BANG score, postoperative analgesic methods, and postoperative SpO₂ and FiO₂ values are recorded, and the SpO₂/FiO₂ ratio is calculated. All data are collected observationally without any additional procedures or changes to standard care.

SUMMARY:
This prospective observational study aims to evaluate the association between postoperative oxygenation, assessed by the SpO₂/FiO₂ ratio, and body mass index (BMI), STOP-BANG score, and postoperative analgesic methods in patients undergoing elective laparoscopic cholecystectomy in the reverse Trendelenburg position. Postoperative SpO₂ and FiO₂ values will be recorded within the first postoperative hour, and the SpO₂/FiO₂ ratio will be calculated. Analgesic techniques applied as part of routine clinical practice will be documented. The study does not involve any additional intervention beyond standard care. The findings are expected to contribute to a better understanding of factors associated with early postoperative oxygenation and hypoxemia risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients who provide written informed consent
* ASA physical status I-III
* Patients undergoing elective laparoscopic cholecystectomy
* Surgery performed in the reverse Trendelenburg position (30°)
* Expected operative duration < 3 hours
* Exclusion Criteria:
* Age < 18 years
* Refusal or inability to provide informed consent
* ASA physical status IV or higher
* Known chronic respiratory diseases (e.g., asthma, COPD)
* Severe cardiac failure (NYHA class III-IV) or advanced cardiovascular disease
* Emergency surgery
* Preoperative oxygen supplementation or baseline SpO₂ < 90%
* Prolonged intubation or perioperative respiratory complications
* Requirement for postoperative noninvasive ventilation or intensive care unit admission
* Missing SpO₂ or FiO₂ data preventing calculation of the SpO₂/FiO₂ ratio

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older with ASA physical status I-III who undergo elective laparoscopic cholecystectomy in the reverse Trendelenburg position. All participants provide written informed consent. Patients with significant respiratory or cardiovascular comorbidities, emergency surgery, or perioperative respiratory complications are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
postoperative SpO₂/FiO₂ Ratio | Within the first postoperative hour (0-60 minutes after surgery)
  The SpO₂/FiO₂ ratio calculated using peripheral oxygen saturation (SpO₂) and fraction of inspired oxygen (FiO₂) measured during the early postoperative period to assess postoperative oxygenation.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

REFERENCES:
- [Background] Perilli V, Sollazzi L, Bozza P, Modesti C, Chierichini A, Tacchino RM, Ranieri R. The effects of the reverse trendelenburg position on respiratory mechanics and blood gases in morbidly obese patients during bariatric surgery. Anesth Analg. 2000 Dec;91(6):1520-5. doi: 10.1097/00000539-200012000-00041. PMID 11094011
- [Result] Aboseif A, Bedewy A, Nafei M, Hammad R, Amin S. Effect of Intraoperative Lung Recruitment and Transversus Abdominis Plane Block in Laparoscopic Bariatric Surgery on Postoperative Lung Functions: A Randomized Controlled Study. Anesth Pain Med. 2023 Mar 5;13(2):e128440. doi: 10.5812/aapm-128440. eCollection 2023 Apr. PMID 37645008